CLINICAL TRIAL: NCT03199456
Title: A Randomized, Controlled, Post-market Clinical Investigation to Evaluate Zip Surgical Skin Closure Device in Comparison of Using Standard of Care Sutures for Laceration Repair in Pediatrics and Adults in an Accident and Emergency Department
Brief Title: A Randomized Post-market Study to Evaluate Zip Device Compared to Sutures for Laceration Repair in Pediatrics and Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZipLine Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zip-009
Record Dates: First submitted 2017-06-19; First posted 2017-06-27 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Laceration
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Zip Surgical Skin Closure Device group (Experimental): The subjects randomised to this arm will be treated with the Zip device for 10 days (+/-2) days.
  Interventions: Device: Zip surgical skin closure device
- Standard of Care sutures group (Active Comparator): The subjects randomised to this arm will be treated with standard of care sutures for 10 days (+/- 2 days).
  Interventions: Device: Standard of Care sutures

INTERVENTIONS:
Device: Zip surgical skin closure device — Zip surgical skin closure device manufactured by ZipLine Medical, Inc. is a CE-marked, non-invasive, single use device that is designated to provide closure of the skin layer for lacerations or surgical incisions.
  Arms: Zip Surgical Skin Closure Device group
Device: Standard of Care sutures — Standard of Care sutures according to the hospitals current clinical praxis.
  Arms: Standard of Care sutures group

SUMMARY:
The Zip-009 clinical investigation will enroll 26 paediatric and adult subjects requiring laceration repair and fulfilling the eligibility criteria for the clinical investigation. The investigation is designed to evaluate the time and cost savings and the satisfaction and outcomes of the Zip device compared to conventional sutures. The subjects will be randomly assigned at a 1:1 ratio to either the Zip Surgical Skin Closure Device group or the Standard of Care sutures group. The investigation consists of one screening/baseline visits at day 0 where the subject will be treated with either the Zip device or sutures, and thereafter two follow up telephone calls at day 10 and day 30. The Zip device/sutures will be removed prior the first follow up call day 10. The duration of the investigation is estimated to 5 months, including a 4-month recruitment period and 1-month follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Between 4 and above at the time of laceration repair.
2. Require suture closure as standard of care for simple straight wounds on trunk, extremities or face.
3. Low Tension Laceration, e.g. skin can be easily approximated by pinching with fingers.
4. Subject and legal representative(s) (if a pediatric subject) are willing and able to comply with the investigational device removal and meet the follow up requirements.
5. Subject and legal representative(s) (if a pediatric subject) have been informed of the nature, the scope and the relevance of the study.
6. Subject and legal representative(s) (if a pediatric subject) have voluntarily agreed to participation and have duly signed the Informed Consent Form.

Exclusion Criteria:

1. Known personal or familial history of scar hypertrophy.
2. Known or suspected allergies or hypersensitivity to non-latex skin adhesives.
3. Atrophic skin deemed clinically prone to blistering.
4. Wounds that are easily susceptible to infection as a result of exposure to unsanitary conditions ("dirty wounds").
5. Wounds that require deep dermal closure using sutures.
6. Known or suspected mental problems and/or aggressiveness that indicates that the subject might try to remove the device during the treatment period.
7. Ongoing treatment with cytostatic.
8. Known or suspected diagnosis of severe anorexia.
9. Participating in any other clinical investigation.
10. Known health condition that would affect healing in the opinion of the investigator.
11. Any subject that according to the Declaration of Helsinki is deemed unsuitable for study enrolment.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Treatment time | Day 0
  The primary endpoint in this clinical investigation is the mean difference in time to wound closure, for the two treatment methods used. These include total treatment time and duration of period starting from the preparation of procedure until protective wound dressing is applied, and including whether or not anesthesia and/or sedation was used when comparing the Zip Surgical Skin Closure Device and the standard of care closure suturing.

SECONDARY OUTCOMES:
Objective evaluation on photographs using Wound Evaluation Score (WES) | Day 0, Day 10 (+/- 2 days), Day 30 (+/- 2 days)
  Difference in Wound Evaluation Score at 10 days and 30 days post-treatment compare to baseline when comparing scar satisfaction and appearance of the subjects receiving Zip Surgical Skin Closure Device versus Standard of Care closure suturing. The score will be based on digital photographs taken on day 0, day 10 and day 30 and made by an independent panel of blinded physician(s).
Subject satisfaction | Day 30 (+/- 2 days)
  Rate of wound healing satisfaction in subject at 30 days post-treatment when comparing Zip Surgical Skin Closure Device versus Standard of Care closure suturing. The endpoint will utilize a questionnaire for the subject to fill out.
Visual Analog Scale (VAS) for pain | Day 0 and Day 10 (+/- 2 days)
  The level of pain in connection to device application and removal measured by a visual analog scale (VAS) 0-100 mm.

OTHER OUTCOMES:
Incidence and severity of Adverse Events (AEs) | 30 days (+/-2 days)
  The incidence and severity of adverse events associated with the Zip Surgical Skin Closure Device and Standard of Care closure sutures.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Malmquist, M.D., Principal Investigator — Funktionsområde Akutsjukvård Barn Solna, Astrid Lindgrens Barnsjukhus, Karolinska Universitetssjukhuset, 171 76 Stockholm, Sweden
Locations (2):
- Sweden (2):
  - Funktionsområde Akut Huddinge, Akutmottagningen Huddinge, Karolinska Universitetssjukhuset, Huddinge
  - Funktionsområde Akutsjukvård Barn Solna, Astrid Lindgrens Barnsjukhus, Karolinska Universitetssjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No